CLINICAL TRIAL: NCT03208309
Title: Effect of Diacerein in the Metabolic Control of Patients With Diabetes Mellitus Type 2 and Secondary Failure to Metformin
Brief Title: Effect of Diacerein in the Metabolic Control of Patients With DM Type 2 and Secondary Failure to Metformin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ANS Pharma (Industry)
Collaborators: University of Campinas, Brazil (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 072/2011; Parecer CEP072/2011 (Other: CEP FCM UNICAMP)
Record Dates: First submitted 2017-06-27; First posted 2017-07-05 (Actual); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: Complications of Diabetes Mellitus; Diabetes Mellitus; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Complications; Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — diacerein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diacerein (Active Comparator): Diacerein 50 mg immediate release capsule, once daily for the starting 28 days and Diacerein 50 mg immediate release capsule twice a day for the remainder of the study.
  Interventions: Drug: Diacerein
- Placebo (Placebo Comparator): Placebo capsules once a day for the starting 28 days and two times daily for the remainder of the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diacerein
  Arms: Diacerein
Drug: Placebo
  Arms: Placebo

SUMMARY:
Considering that, Diacerein is on the market for 16 years being used continuously in elderly patients with osteoarthritis without experience significant side effects, and considering the anti-hyperglycemic effect and the improvement in the insulin resistance observed in animal models of type 2 diabetes treated with this medicine.

The aim of this study is to investigate the effect of Diacerein, a medication with anti-osteoarthritic properties and moderately analgesic activity, anti-inflammatory and antipyretic, which demonstrates inhibit properties for the synthesis of pro-inflammatory cytokines such as interleukin 1 (IL-1). Administered for 12 weeks and the effect in the glycemic and metabolic control in patients with diabetes mellitus 2 and secondary failure to metformin treatment.

DETAILED DESCRIPTION:
This proof of concept study aims to access the metabolic control in patients with type 2 diabetes mellitus and secondary failure to metformin.

The Study is a Phase II, Multicenter, National, Prospective, Randomized, Double-blind, Parallel Groups, Placebo Comparative Trial. UNICAMP (Hospital of Unicamp) is the coordinator center and the investigators and research center participating are from the State University of Feira de Santana (BA) and the Center for Diabetes and Hypertension in Fortaleza (CE).

Study Objectives: To investigate the effect of Diacerein administered for 12 weeks; glycemic and metabolic control; in patients with diabetes mellitus type 2 and secondary failure to metformin treatment. The Total Number of patients will be approximately 60, 30 patients in each group.

Diagnostic Criteria - Diabetes mellitus type 2 between 6 months to 10 years of disease, body mass index between 25 and 35 kg/m2, fasting glucose between 120 and 250 mg / dL, glycated Hb A1c greater than 7,5 % and taking metformin (dose above 1700 mg / day) with or without other secretagogue.

Inclusion Criteria - male or female (not pregnant) , aged between 35 and 65 years who present clinical symptoms of type 2 diabetes between 6 months to 10 years of disease, according to the diagnostic criteria.

Exclusion Criteria - Patients with DM1, DM2 using insulin and other types of diabetes.

T2DM with chronic complications that already have clinical consequences, serum creatinine greater than 1.5 mg/dl, history of heart disease and severe concomitant diseases such as liver, coronary artery, renal, with severe psychiatric or neurological disorders .

Patients with a history of abuse of alcohol and / or illegal drugs or psychotropic medicines in the past six months, hypersensitivity to any of the components of the of study drug formulation.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus type 2 between 6 months to 10 years of disease
* Body mass index between 25 and 35 kg/m2
* Fasting glucose between 120 and 250 mg / dL
* Glycated Hb A1c greater than 7,5 % and taking metformin (dose above 1700 mg / day) with or without other secretagogue
* Male or female (not pregnant), who present clinical symptoms of type 2 diabetes between 6 months to 10 years of disease, according to the diagnostic criteria.

Exclusion Criteria:

* Patients with DM1, DM2 using insulin and other types of diabetes
* T2DM with chronic complications that already have clinical consequences
* Creatinine serum greater than 1.4 (female) and 1.5 mg/dl (male)
* History of heart disease and severe concomitant diseases such as liver, coronary artery, renal, with severe psychiatric or neurological disorders
* Patients with a history of abuse of alcohol and/or illegal drugs or psychotropic medicines in the past six months
* Hypersensitivity to any component of the of study drug and placebo formulation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Fasting Glucose | 4 weeks
HbA1c - glycated haemoglobin | 12 weeks
Cholesterol | 12 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- Brazil (3):
  - Centro de Estudos em Diabetes e Hipertensão, Fortaleza, Ceará
  - Universidade Estadual de Feira de Santana, Feira de Santana, Estado de Bahia
  - Universidade Estadual de Campinas, Campinas, São Paulo

REFERENCES:
- [Background] Ramos-Zavala MG, Gonzalez-Ortiz M, Martinez-Abundis E, Robles-Cervantes JA, Gonzalez-Lopez R, Santiago-Hernandez NJ. Effect of diacerein on insulin secretion and metabolic control in drug-naive patients with type 2 diabetes: a randomized clinical trial. Diabetes Care. 2011 Jul;34(7):1591-4. doi: 10.2337/dc11-0357. Epub 2011 May 24. PMID 21610123
- [Background] Velloso LA, Folli F, Perego L, Saad MJ. The multi-faceted cross-talk between the insulin and angiotensin II signaling systems. Diabetes Metab Res Rev. 2006 Mar-Apr;22(2):98-107. doi: 10.1002/dmrr.611. PMID 16389635
- [Background] Tobar N, Oliveira AG, Guadagnini D, Bagarolli RA, Rocha GZ, Araujo TG, Prada PO, Saad MJ. Comment on: Ramos-Zavala et al. Effect of diacerein on insulin secretion and metabolic control in drug-naive patients with type 2 diabetes: a randomized clinical trial. Diabetes Care 2011;34:1591-1594. Diabetes Care. 2012 Feb;35(2):e13; author reply e14. doi: 10.2337/dc11-1856. No abstract available. PMID 22275450
- [Background] Tobar N, Oliveira AG, Guadagnini D, Bagarolli RA, Rocha GZ, Araujo TG, Santos-Silva JC, Zollner RL, Boechat LH, Carvalheira JB, Prada PO, Saad MJ. Diacerhein improves glucose tolerance and insulin sensitivity in mice on a high-fat diet. Endocrinology. 2011 Nov;152(11):4080-93. doi: 10.1210/en.2011-0249. Epub 2011 Sep 6. PMID 21896669